CLINICAL TRIAL: NCT06106061
Title: Effectiveness and Safety of the Facet Fixation (FFX®) Implant in the Treatment of Degenerative Lumbar Spinal Stenosis
Acronym: FFX® RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SC Medica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-A01382-43
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Degenerative Lumbar Spinal Stenosis
MeSH Terms: interventions — Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one: Decompression + FFX® (Experimental)
  Interventions: Device: Decompression + FFX®
- Group two: Decompression alone (Active Comparator)
  Interventions: Procedure: Decompression alone

INTERVENTIONS:
Device: Decompression + FFX® — Surgical treatment of degenerative lumbar spinal stenosis by spinal decompression associated with the use of FFX® implant
  Arms: Group one: Decompression + FFX®
Procedure: Decompression alone — Surgical treatment of degenerative lumbar spinal stenosis by spinal decompression alone
  Arms: Group two: Decompression alone

SUMMARY:
This is a prospective, multicentric, comparative, randomised-controlled study to evaluate the safety and efficacy of the Facet Fixation implant.

The main objective is to evaluate the effectiveness of spinal decompression associated with FFX® implants compared to spinal decompression alone in treating lumbar spinal stenosis after 2 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years.
* Radiographic confirmation of clinical symptoms of at least moderate degenerative spinal stenosis, of 1 to 3 adjacent segments in the L1-S1 region with the need for surgical decompression.
* Radiographic confirmation of no translational instability in main segment as well as in adjacent segments (dynamic translational instability ≤3 mm);
* Visual analogue scale (VAS) back pain score ≥ 50 mm (on a 100-mm scale).
* Minimum of 3 months of conservative therapy without improvement of symptoms.
* Mental & physical ability of the subject to follow the protocol (i.e., compliance with time schedule & treatment plan, able to fill in questionnaire & to undergo further study procedures).
* Personally signed and dated informed consent document prior to any study-related procedures indicating that the subject has been informed of all pertinent aspects of the clinical investigation.

Exclusion Criteria:

* Prior lumbar spine surgery.
* Radiographically confirmed damage of a vertebral body (e.g., osteoporotic compression fracture or because of tumours), at any lumbar level.
* Isthmic or degenerative spondylolisthesis (anterolisthesis; retrolisthesis ≥ grade II) or spondylolysis (pars fracture).
* Degenerative lumbar scoliosis (Cobb angle > 25°).
* Adipositas (obesity); defined as a body mass index (BMI) >40.
* Pregnancy, or wish to get pregnant during the course of the study, or breastfeeding.
* Known allergy or sensitivity to titanium, titanium alloys, or MRI contrast agents.
* Active or chronic infection-systemic or local.
* History of significant peripheral neuropathy.
* Significant peripheral vascular disease (e.g., with diminished dorsalis pedis or posterior tibial pulses).
* Paget disease, osteomalacia or other metabolic bone disorders.
* Cauda equina syndrome.
* Known or documented history of transmissible disease, including AIDS, HIV and active hepatitis.
* More than 3 vertebral levels requiring surgery.
* Disc herniation at any lumbar level requiring surgical intervention.
* Known osteoporosis (bone mineral density, BMD < 120 mg/cm3).
* Chronically taking medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., steroids), not including a Medrol (methylprednisolone) dose pack.
* Fixed and complete motor, sensory, or reflex deficit.
* Rheumatoid arthritis or other autoimmune diseases.
* Active malignancy: a subject with a history of any invasive malignancy (except non-melanoma skin cancer) unless he/she has been treated with curative intent and there has been no clinical signs or symptoms of the malignancy for at least 5 years. Subjects with a primary bony tumour are excluded as well.
* Subject with a history of substance abuse (e.g., recreational drugs, narcotics, or alcohol).
* Bone destruction, demineralisation or any affection potentially affecting fixation of an implant.
* Spondylodiscitis or spine tumour.
* Currently seeking or receiving workman's compensation.
* In active spinal litigation.
* Subjects who participate(d) in another clinical trial (within the last 4 weeks) that might influence the safety & effectiveness assessment of this trial.
* Subjects who are lawfully kept in an institution.
* Subject who, in the opinion of the investigator, will be inappropriate for inclusion in this clinical trial or who will not comply with requirements of the study.
* Subject under supervision or legal guardianship, or judicial protection.
* Subject deprived of liberty by judicial or administrative decision.
* Subject not covered by a social security scheme.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with composite clinical success (CCS) | 2 years
  The CCS will be considered as met if ALL of the following criteria are satisfied for a subject:
  * Back pain score (VAS) decrease by more than 20 mm (on 100-mm scale)
  * No secondary surgical intervention at the index level (excluding wound problems)
  * No non-surgical lumbar treatment of interest at any lumbar level